CLINICAL TRIAL: NCT00002676
Title: PHASE II TRIAL OF CHEMOTHERAPY PLUS RADIOTHERAPY FOR MANAGEMENT OF PRIMARY CENTRAL NERVOUS SYSTEM NON-HODGKIN'S LYMPHOMA (PCNSL)
Brief Title: Chemotherapy and Whole-Brain Radiation Therapy in Treating Patients With Primary Central Nervous System Non- Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-937351; E-N9371; CDR0000064319 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHOD + BVAM + WBRT (Experimental): Patients 70 years old and younger with newly diagnosed, biopsy-proven PCNSL received one cycle of CHOD followed by two cycles of BVAM. Patients then received WBRT, 30.6 Gy, if a complete response was evoked, or 50.4 Gy if the response was less than complete; both doses were given in 1.8-Gy daily fractions.
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells and may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and whole-brain radiation therapy in patients with primary central nervous system non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response to CHOD (cyclophosphamide/doxorubicin/vincristine/ dexamethasone) and BVAM (carmustine/vincristine/cytarabine/methotrexate) plus whole-brain radiotherapy in patients with primary central nervous system non-Hodgkin's lymphoma (PCNSL). II. Assess the toxic effects associated with this treatment. III. Assess the survival of patients with PCNSL receiving this treatment. IV. Investigate the frequency of systemic involvement at follow-up. V. Identify factors that appear to be associated with outcome.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary central nervous system non-Hodgkin's lymphoma (PCNSL) Clinically diagnosed intracranial space-occupying lesion Pathology consistent with non-Hodgkin's lymphoma and reviewed by NCCTG Biopsy optional if characteristic history, pathognomonic neuroimaging, and cytology are consistent with malignant lymphocytes from vitrectomy, CSF, or both No occult systemic lymphoma or prior lymphoma No post-transplant lymphoproliferative disorder Disease measurable or evaluable on postoperative contrast-enhanced CT or MRI Postoperative therapy must start within 6 weeks of definitive diagnosis

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: ECOG 0-3 Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 120,000/mm3 Hepatic: Bilirubin no greater than 2 times normal AST no greater than 2 times normal Renal: Creatinine no greater than 1.5 times normal Cardiovascular: No heart failure No uncontrolled arrhythmia Pulmonary: No severe pulmonary failure Other: No serious uncontrolled infection No active bleeding No AIDS or HIV-positive serology No prior organ transplant No pregnant or nursing women Negative pregnancy test required of fertile women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Corticosteroids allowed if dose fixed or decreasing for at least 1 week prior to baseline scan Radiotherapy: No prior radiotherapy Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1995-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 10 years

SECONDARY OUTCOMES:
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. O'Neill, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (21):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Laack NN, O'Neill BP, Ballman KV, O'Fallon JR, Carrero XW, Kurtin PJ, Scheithauer BW, Brown PD, Habermann TM, Colgan JP, Gilbert MR, Hawkins RB, Morton RF, Windschitl HE, Fitch TR, Pajon ER Jr; North Central Cancer Treatment Group and Mayo Clinic. CHOD/BVAM chemotherapy and whole-brain radiotherapy for newly diagnosed primary central nervous system lymphoma. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):476-82. doi: 10.1016/j.ijrobp.2010.06.002. Epub 2010 Aug 26. PMID 20800387
- [Result] O'Neill BP, O'Fallon JR, Cha SS, et al.: Newly diagnosed primary central nervous system lymphoma (PCNSL): initial report of North Central Cancer Treatment Group (NCCTG)/Eastern Cooperative Oncology Group (ECOG) protocol 93 73 51. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2074, 2002.